CLINICAL TRIAL: NCT07052344
Title: Gut-Brain Neural Coupling in Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Gary Farkas, Assistant Professor, University of Miami
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 20250237
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: SCI - Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-load Condition Meal Group (Experimental): Participants will be in this group for up to 2 weeks.
  Interventions: Other: Preload condition; Other: Ad-libitum control condition
- Ad-libitum Condition Meal Group (Active Comparator): Participants will be in this group for up to 2 weeks.
  Interventions: Other: Ad-libitum control condition

INTERVENTIONS:
Other: Preload condition — Participants will consume a fixed compulsory preload meal of Campbell's Tomato soup (~300 grams) 30 minutes after the baseline assessments. Fifteen minutes after consuming the preload meal, participants will receive the ad libitum test meal, consisting of a pre-weighed serving of Stouffer's Macaroni and Cheese (~700 g).The pre-load condition will be completed at only one of two visits. Participation will be up to 2 weeks with the visits separated by up to 2 weeks. Duration for the pre-load condition visit will be up to 6 hours
  Arms: Pre-load Condition Meal Group
Other: Ad-libitum control condition — Participants will only consume the ad libitum test meal, which consists of a pre-weighted serving of Stouffer's Macaroni and Cheese (~700 g). The ad-libitum meal will be consumed at both visits. Participation will be up to 2 weeks with the visits separated by up to 2 weeks. The ad-libitum control condition visit will take up to 2 hours.

SUMMARY:
The purpose of this research is to determine the effects of food on brain and stomach activity in persons with and without spinal cord injury (SCI).

ELIGIBILITY:
Inclusion Criteria, SCI and Controls

* Adults, 18 to 70 years of age.
* Sex, male or female.
* Weight-stable (±3 kg) for the preceding 3 months (self-report).
* Physically inactive adults not meeting weekly activity guidelines (<150 min/week) for the preceding 3 months (self-report).
* Fluent in written and spoken English.

Exclusion Criteria, SCI and Controls

* Do not meet the inclusion criteria.
* Current/regular smoker (defined by Center for Disease Control (CDC)/ National Institute of Health (NIH) as an adult who has smoked 100 cigarettes in his or her lifetime and who currently smokes either every day or every other day) (self-report).
* Currently dieting and/or trying to gain or lose weight.
* Vagus or recurrent laryngeal nerve injury (self-report).
* Uncontrolled thyroid disease, such that they are not on thyroid medication (e.g., levothyroxine) to treat the condition (self-report)
* Diabetes (type 1 or type 2) and/or currently taking anti-diabetic or glucagon-like peptide-1 (GLP-1)/dual agonist medications (self-report).
* Gastrointestinal disease (self-report), such as inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis), celiac disease, irritable bowel syndrome, gastroesophageal reflux disease, peptic ulcer disease, chronic pancreatitis, liver cirrhosis, and any condition requiring gastrointestinal surgery (e.g., bowel resection, colostomy, or ileostomy).
* Swallowing disorder (self-report).
* History of bariatric surgery
* Food allergies/dislikes or dietary restrictions (i.e. vegan) (self-report).
* Allergy to adhesives (self-report)
* Open abdominal wounds or abdominal skin not intact.
* Current use of probiotics/prebiotics (self-report).
* Current use of medications that can impact appetite, body weight, and/or bowel function, such as prokinetic, antiemetic, narcotic analgesics, anticholinergic, anti-inflammatory, antipsychotic, or anti-obesity agents (self-report).
* Pregnant (determined by urine pregnancy test) or breastfeeding women.
* Non-adults (infants, children, teenagers).
* Adults unable to consent
* Prisoner.

SCI-specific Eligibility Criteria

Inclusion Criteria, SCI Only

* At least 12 months post-SCI, denoting chronic injury
* Complete American Spinal Injury Association (ASIA) Impairment Scale (AIS A) or motor-incomplete (AIS B) tetraplegia (SCI at or above C8 lesion)
* Able to self-feed (self-report)
* On a bowel care program every day or every other day (self-report).

Exclusion Criteria, SCI Only

* Under 12 months post-SCI.
* Motor-incomplete (AIS C, D) paraplegia (SCI below C8 lesion), including thoracic, lumbar, and sacral injuries.
* Ventilator-dependence (self-report).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase amplitude coupling (PAC) strength | up to 2 weeks
  Gut-brain connectivity will be assessed using phase-amplitude coupling (PAC) to examine the interaction between gastric electrical oscillations and cortical rhythms. PAC will be calculated from electrophysiological raw data to produce one unitless value ranging from -1 to 1, for each subject. The higher the value, the greater the gut-brain connectivity/PAC strength.

CONTACTS AND LOCATIONS:
Overall Officials: Gary J Farkas, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami - Miami Project to Cure Paralysis, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No